CLINICAL TRIAL: NCT03029728
Title: Biomarker for Hereditary AngioEdema Disease: An International, Multicenter, Longitudinal Monitoring Protocol
Brief Title: Biomarker for Hereditary AngioEdema Disease
Acronym: BioHAE
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BHAE 06-2018
Record Dates: First submitted 2017-01-18; First posted 2017-01-24 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2021-03

CONDITIONS: C1 Esterase Inhibitor Deficiency; Angio Edema; C4 Deficiency; HAE; Hereditary Angioedema; Hereditary Angioedema Type II; Hereditary Angioedema Type III; Hereditary Angioedema Type I
Keywords: Hereditary Angioedema; Biomarker; Hereditary Angioedema Type I; Hereditary Angioedema Type II; Hereditary Angioedema Type III
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema; Hereditary Angioedema Types I and II; Hereditary Angioedema Type III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Hereditary Angioedema: Participants diagnosed with Hereditary Angioedema disease aged between 2 months and 60 years

SUMMARY:
International, multicenter, observational, longitudinal monitoring study to identify, validate and/or monitor Mass Spectrometry (MS)-based biomarker/s for Hereditary Angioedeme (HAE) disease and to test the clinical robustness, specificity, and predictive value of theese biomarker/s

DETAILED DESCRIPTION:
Hereditary Angioedema (HAE) is a rare autosomal dominant genetic disorder, characterized by recurrent episodes of angioedema of the face, larynx, lips, abdomen, and extremities.The most common types of HAE develop as result of mutations in the SERPING1 gene that encodes the C1 inhibitor (C1-INH), a protease involved in limiting bradykinin production. Excessive bradykinin due to low levels of C1-INH (HAE type 1) or dysfunctional C1-INH (HAE type 2) leads to capillary leakage and angioedema formation. The third type of HAE is not associated with a C1-INH deficiency, develops as a result of mutations in the Factor 12 gene (FXII) and affects almost exclusively women. Rare cases of HAE have also been described resulting from mutations in Plasminogen (PLG), Angiopoetin 1 (ANGPT1), and Kininogen 1 (KNG1).

The characteristic symptom of hereditary angioedema is recurrent episodes of swelling due to the accumulation of excessive body fluid. The most commonly affected areas of the body include the hands, feet, eyelids, lips, genitals, larynx and gastrointestinal tract. The most serious complication of HAE is laryngeal edema that can become life threatening; but it is a relatively rare event.

The diagnosis of hereditary angioedema is made by a thorough clinical evaluation, a detailed patient history, and blood tests.Clinical diagnosis is complicated because HAE is highly variable in the clinical phenotype and the majority of the physicians believe that they never seen a patient with that disorder. Laboratory diagnosis involves measurement of the C1-INH function, C1-INH and C4 levels. Both C1-INH protein level and function is low in HAE-1 patients, whereas in HAE-2 individuals the C1-INH concentrations is optimal or even elevated, however C1-INH function is impaired. Generally, C4 levels are low in both HAE-1/2 patients.

CENTOGENE utilizes Liquid Chromatography-Multiple Reaction Monitoring Mass Spectrometry (LC-MRM-MS) method to identify potential disease-specific biomarkers for HAE. Such biomarker/s may support the early diagnosis and treatment monitoring and personalization in the future.

Therefore, it is the goal of this study is to identify new biomarkers for HAE, validate the identified biomarkers, and monitor these biomarkers longitudinally to determine their clinical robustness, specificity, and predictive value.

ELIGIBILITY:
INCLUSION CRITERIA

* Informed consent is obtained from the participant or participant's parent/legal guardian
* The participant is aged between 2 months and 60 years
* The diagnosis of Hereditary Angioedema is confirmed by CENTOGENE

EXCLUSION CRITERIA

* Inability to provide informed consent
* Participant is younger than 2 months or older than 60 years
* The diagnosis of Hereditary Angioedema disease is not confirmed by CENTOGENE

Ages: 2 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants diagnosed with Hereditary Angioedema (HAE) disease
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Identification, validation and/or monitoring of mass spectrometry (MS)-based biomarkers of Hereditary Angioedema (HAE) patients | 36 months
  All samples will be analyzed for the identification of biomarker/s via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

SECONDARY OUTCOMES:
Determination of the clinical robustness, specificity, and predictive value of the biomarker(s) | 36 months
  Samples will be analyzed for the identified biomarker candidates via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, MD, Study Chair — CENTOGENE GmbH
Locations (7):
- Arabkir JMC-ICAH, Yerevan, Armenia
- Center of Allergy and Immunology, Tbilisi, Georgia
- Department of Pediatric Genetics, Amrita Institute of Medical Sciences & Research Centre, Kerola, India
- Clinica San Pablo de Surco, Lima, Peru
- Szpital Uniwersytecki w Krakowie, Krakow, Poland
- Centrul Clinic Mediquest, Târgu Mureş, Romania
- Sakarya University Research and Training Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided